CLINICAL TRIAL: NCT06572462
Title: Application of Thymoglobulin (ATG) Individualized Dosing Model in Unrelated Allogeneic Hematopoietic Stem Cell Transplantation.
Brief Title: ATG Individualized Dosing Model in URD-PBSCT.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2023-794-01
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Cytomegalovirus Infections; Infection Reactivation; Stem Cell Transplant Complications
MeSH Terms: conditions — Cytomegalovirus Infections; Latent Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- targeted dosing ATG cohort (Experimental): The targeted dosing ATG cohort received the same dose of medication at -5 days and -4 days as the traditional administration method (-5days, 1.5mg/kg; -4days 2.5mg/kg), Two individual doses were given on -3days and day -2days according to the dose adjustment strategy.
  Interventions: Drug: individualized ATG dosing strategy

INTERVENTIONS:
Drug: individualized ATG dosing strategy — Investigators quantified active ATG exposure in 106 haploidentical peripheral blood stem cell transplantation (haplo-PBSCT) recipients, who received a conventional fixed dose of 10 mg/kg ATG during conditioning, the optimal concentration range of active ATG-AUC was determined through the application of machine learning methods, was found to be 100-148.5 × 10^3 UE·d/L. This concentration range was associated with a reduction in CMV/EBV reactivation, without an increase in acute GVHD or malignant disease relapse. Mathematical function was then exploited to determine the total targeted ATG dose on -3days to -2days based on concentrations of active ATG on -5daysto -4days. Based on this function, investigators established a dosing strategy that aimed to maintain the active ATG-AUC within the optimal range.

SUMMARY:
Anti-thymocyte globulin (ATG) is widely used in allogeneic hematopoietic stem cell transplantation to prevent severe graft-versus-host disease (GVHD) and graft failure. However, overexposure to ATG may increase cytomegalovirus (CMV), Epstein-Barr virus (EBV) reactivation, non-relapse mortality, and disease recurrence. A targeted dosing strategy was established based on ATG concentration monitoring and conducted a phase 2 trial to evaluate the safety and efficacy of the dosing strategy in adult unmanipulated haplo-PBSCT, a encouraging result was attained. In this trial, The ATG-targeted dosing strategy was extended to adult unrelated donor allogeneic hematopoietic stem cell transplantation, ATG was administered for 4 days (-5 days to -2 days) during conditioning. The ATG doses on-3 days and- 2days were adjusted by our dosing strategy to achieve the optimal ATG exposure. The primary endpoint was CMV reactivation on +180 days.

DETAILED DESCRIPTION:
Allogeneic hematopoietic cell transplantation(allo-HCT) is a curative therapy for hematological disorders and the ATG is commonly used as prophylaxis for GVHD. Previous studies have indicated that there is an optimal dosage for ATG administration, if the dosage is too high, it may affect engraftment and increase the risk of infection and relapse, whereas an inadequate dosage may increase the risk of acute or chronic GVHD, there is still controversy about the optimal dose of ATG, its pharmacologic effects on clinical outcomes of HSCT are associated with donor source, human leukocyte antigen (HLA) disparity, conditioning intensity, and GVHD prophylaxis, so although has been investigated for decades, the optimal dosage of ATG in allogeneic hematopoietic stem cell transplantation remains undetermined.

ATG exerts pharmacologic effects in its active form upon binding to lymphocytes, and its exposure is presented as the area under the concentration-time curve (AUC). To obtain plasma active ATG concentrations, investigators developed an active ATG concentration detection method based on flow-cytometry with HUT-78 T-cells. In previous study, investigators quantified active ATG exposure in 106 haploidentical peripheral blood stem cell transplantation (haplo-PBSCT) recipients, who received a conventional fixed dose of 10 mg/kg ATG during conditioning, the optimal concentration range of active ATG-AUC was determined through the application of machine learning methods, was found to be 100-148.5 × 10^3 UE·d/L. This concentration range was associated with a reduction in CMV/EBV reactivation, without an increase in acute GVHD or malignant disease relapse. Mathematical function was then exploited to determine the total targeted ATG dose on -3days to -2days based on concentrations of active ATG on -5daysto -4days. Based on this function, a dosing strategy was established that aimed to maintain the active ATG-AUC within the optimal range. To validate this individualized dosing strategy, investigators conducted a single-arm, phase 2 trial, demonstrating that this strategy could reduce CMV/EBV reactivation and improve survival without increasing the incidence of GVHD after haplo-PBSCT. Given the similarity between unrelated donor hematopoietic stem cell transplantation (URD-HSCT) and haploidentical hematopoietic stem cell transplantation (haplo-HSCT) in terms of conditioning regimens, GVHD prophylaxis, and supportive therapies, as well as the conventional fixed dose of 10mg/kg employed in both settings, investigators have designed and conducted a single-center, prospective, single-arm clinical trial. The aim of this trial is to translate the individualized ATG dosing strategy, which was originally developed based on ATG concentration monitoring in haplo-HSCT patients, to URD-HSCT, with the goal of further validating its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant hematological tumors who have indications for allogeneic hematopoietic stem cell transplantation.
2. HLA-matched unrelated donor
3. Patient age ≥14 years old and ≤65 years old
4. ALT and AST ≤ 2.5 times the upper limit of normal values, bilirubin ≤ 2 times the upper limit of normal values
5. Creatinine ≤ high limit of normal value
6. No uncontrollable infection or serious mental illness
7. Physical strength score is 0-2 (ECOG)
8. Sign the informed consent form

Exclusion Criteria:

1. Unrelated donor who is not HLA matched
2. No indication for allogeneic hematopoietic stem cell transplantation
3. Patient age <14 years old or >65 years old
4. The donor or recipient are pregnant
5. Suffering from mental illness or other conditions and being unable to proceed as planned

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of CMV reactivation | 0Day-180Days
  The primary endpoint was the cumulative incidence of CMV reactivation on +180 days after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: diahong Liu, MD, Principal Investigator — First Medical Center of Chinese PLA General Hospital
Locations (1):
- Department of Hematology, First Medical Center of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen S, Wang L, Luan S, Wang H, Du J, Ge D, Li F, Wu Y, Gu Z, Dou L, Liu D. Reduced cytomegalovirus reactivation and viremia without increasing GVHD after URD-PBSCT: A prospective study using targeted ATG dosing strategy. Cancer Pathog Ther. 2025 Apr 5;4(2):145-152. doi: 10.1016/j.cpt.2025.04.001. eCollection 2026 Mar. PMID 41624481